CLINICAL TRIAL: NCT06335589
Title: Adapting Treatment Delivery to Improve Retention in Evidence-Based PTSD Treatment (CDA 21-191)
Brief Title: Adapting Treatment Delivery to Improve Retention in Evidence-Based PTSD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDX 24-002
Record Dates: First submitted 2024-03-06; First posted 2024-03-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Psychotherapy; Mental Health; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Massed PTSD treatment (e.g., cognitive processing therapy [CPT] or prolonged exposure [PE] therapy delivered at least 3 times per week) will be compared to CPT & PE delivered as usual, which is usually once per week.
Who Masked: Outcomes Assessor
Masking Description: Clinical interviewers who assess primary outcomes will not be informed of participant's randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBP-Massed (Experimental): PTSD evidence-based psychotherapies are delivered in a massed format (e.g., intended be delivered at least three times per week).
  Interventions: Other: EBP-Massed
- EBP-TAU (Active Comparator): PTSD evidence-based psychotherapies are delivered treatment as usual, which is typically once per week.
  Interventions: Other: EBP-TAU

INTERVENTIONS:
Other: EBP-Massed — CPT or PE will be delivered in a massed format (e.g., sessions at least 3 days per week)
  Arms: EBP-Massed
Other: EBP-TAU — CPT or PE will be delivered treatment as usual, which is typically once per week.
  Arms: EBP-TAU

SUMMARY:
Posttraumatic stress disorder (PTSD) is prevalent among Veterans and effective evidence-based psychotherapies (EBPs) for PTSD have been implemented within the Veterans Health Administration (VHA). However, retention in PTSD EBPs is poor. Premature dropout is associated with worse clinical outcomes and greater healthcare utilization. Delivery of PTSD EBPs in a massed format, typically three or more days per week delivered within a month, have shown promise for increasing retention. The present study is a pilot feasibility and acceptability study comparing massed PTSD treatment to treatment as usual (e.g., typically weekly treatment).

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 18 years or older;
* meets criteria for current PTSD;
* willingness to be randomized to either condition (e.g., EBP-Massed or EBP-TAU);
* decision to receive CPT or PE in a treatment planning session with a Durham Trauma Recovery Program clinic provider;
* ability to provide informed consent

Exclusion Criteria:

* High acute suicide risk;
* active manic symptoms that would likely interfere with treatment;
* active psychotic symptoms that would likely interfere with treatment;
* currently in a concurrent trauma-focused evidence-based treatment for PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Treatment completion | Immediately after treatment completion or discontinuation (weeks 0-20)
  Proportion of Veterans who complete a full course of an assigned PTSD treatment
Acceptability of Intervention (AIM) | Immediately after treatment completion or discontinuation (weeks 0-20)
  Veterans' perceived acceptability of massed treatment for PTSD; scale score ranges from 1-5; greater score = greater acceptability
Client Satisfaction Questionnaire-8 (CSQ-8) | Post-treatment (weeks 0-20)
  Veterans' perceived satisfaction of assigned treatment; range 8-32; greater scores = greater satisfaction
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Severity Score | Post-treatment (weeks 0-20)
  PTSD Symptom Severity - Clinician Assessed; range 0-80; higher scores = greater severity.
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Severity Score | 3 Month Follow up
  PTSD Symptom Severity - Clinician Assessed; range 0-80; higher scores = greater severity.

SECONDARY OUTCOMES:
Session attendance | Post-treatment (weeks 0-20)
  The number of sessions attended of the assigned treatment
Patient Health Questionnaire-9 (PHQ-9) | Post-treatment (weeks 0-20)
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Patient Health Questionnaire-9 (PHQ-9) | 3 Month Follow Up
  Self-reported depression; range = 0-27; higher scores = more severe symptoms
Brief Inventory of Psychosocial Functioning (BIPF) | Post-treatment (weeks 0-20)
  PTSD-related psychosocial functioning; higher scores = more functional impairment. Items are scored on a Likert scale from 0 (never) to 6 (always). Participants are instructed to skip any item that does not reflect a domain that they have participated in over the past 30 days. The B-IPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100.
Brief Inventory of Psychosocial Functioning (BIPF) | 3 Month Follow up
  PTSD-related psychosocial functioning; higher scores = more functional impairment. Items are scored on a Likert scale from 0 (never) to 6 (always). Participants are instructed to skip any item that does not reflect a domain that they have participated in over the past 30 days. The B-IPF is scored by summing the scored items to create a total score, dividing the total score by the maximum possible score based on the number of items scored, and multiplying by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Y Wells, PhD MS BA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT06335589/ICF_000.pdf